CLINICAL TRIAL: NCT00578539
Title: T-Regulatory Cell Kinetics for Patients Receiving Alemtuzamb and Undergoing Stem Cell Transplantation From HLA Mismatched-Related, or HLA Matched, or One Antigen Mismatched-Unrelated Donors
Brief Title: T-Reg Cell Kinetics, Stem Cell Transplant, REGALE
Acronym: REGALE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-21079-REGALE; REGALE; NCT00647010 (obsolete NCT alias)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Leukemia; Hodgkin Lymphoma; Non Hodgkin Lymphoma; Myeloproliferative Disorders
Keywords: Stem Cell Transplantation
MeSH Terms: conditions — Leukemia; Hodgkin Disease; Lymphoma, Non-Hodgkin; Myeloproliferative Disorders | interventions — Cytarabine; Cyclophosphamide; Mesna; Whole-Body Irradiation; Radiation; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell Transplant (Experimental): All patients will receive Ara C IV every 12 hours for 6 doses starting at 1400 hours on day -8. Cyclophosphamide IV once daily on day -7 and day -6 starting at 1400 hours. MESNA will be administered 15 minutes prior to each dose of Cyclophosphamide and 3, 6, 9, and 12 hours after each dose of Cyclophosphamide. Campath 1h will be given on day -4, day -3, day -2 and day-1. TBI (Total Body Irradiation) will be delivered in 8 fractions of 1.75 Gy in two fractions on day -4, day -3, day -2, and day -1. Stem cell Infusion are infused on day 0.
  Interventions: Drug: ARA C; Drug: Cyclophosphamide; Drug: MESNA; Radiation: Total Body Irradiation (TBI); Biological: Campath-1h; Procedure: Stem Cell Infusion

INTERVENTIONS:
Drug: ARA C — Ara C (3000 mg/m2) IV every 12 hours for 6 doses (days -8 to -5)
  Other Names: Cytarabine
Drug: Cyclophosphamide — Cyclophosphamide (45mg/kg) IV once daily on day -7 and day -6
  Other Names: Cytoxan
Drug: MESNA — MESNA (45mg/kg; divided into 5 doses) will be administered 15 minutes prior to each dose of Cyclophosphamide and 3, 6, 9, and 12 hours after each dose of Cyclophosphamide.
  Other Names: Mesnex
Radiation: Total Body Irradiation (TBI) — TBI: total dose 14.0 Gy, will be delivered in 8 fractions of 1.75 Gy in two fractions on day -4, day -3, day -2, and day -1
  Other Names: Radiation
Biological: Campath-1h — CAMPATH (3 mg IV for patients between 5 and 15 kg; 5 mg for patients between 16 and 30 kg; and 10 mg for patients greater than 30 kg) will be given on day -4, day -3, day -2 and day-1.
  Other Names: Alemtuzumab
Procedure: Stem Cell Infusion — Stem cells are infused on day 0

SUMMARY:
Patients have a type of blood cell disorder that is very hard to cure. We are now suggesting a treatment that might help patients live longer without disease than other treatment plans would. This treatment is known as a stem cell transplant. We believe this may help patients as it allows us to give much stronger doses of drugs and radiation to kill the diseased cells than we could give without the transplant. We also think that the healthy cells may help fight any diseased cells left after the transplant.

Stem Cells are special "mother" cells that are found in the bone marrow (the spongy tissue inside bones), although some are also found in the bloodstream (peripheral blood). As they grow, they become either white blood cells which fight infection, red blood cells which carry oxygen and remove waste products from the organs and tissues or platelets, which enable the blood to clot. For the transplant to take place, we will collect these stem cells from a "donor" (a person who agrees to donate these cells) and give them to recipient. Patients do not have a sibling that is a perfect match, so the stem cells will come from a donor who is the best match available. This person may be a close relative or an unrelated person whose stem cells best "matches" the patients, and who agrees to donate stem cells. Before the transplant, two very strong drugs plus total body irradiation will be given to the patient (pre-conditioning). This treatment will kill most of the blood-forming cells in the bone marrow. We will then give the patient the healthy stem cells. Once these healthy stem cells are in the bloodstream they will move to the bone marrow (graft) and begin producing blood cells that will eventually mature into healthy red blood cells, white blood cells and platelets.

This research study will also use CAMPATH-1H as a pre-treatment. CAMPATH-1H is an antibody against certain types of blood cells. CAMPATH-1H is important because it stays active in the body for a long time after infusion, which means it may work longer at preventing GvHD symptoms.

The stem cell transplant described above is considered to be "standard" treatment. We would like to collect additional blood as described below in order to evaluate how the immune system is recovering.

We are asking permission to draw blood from the patient so that we can measure the number of certain blood cells called T regulatory cells. T regulatory cells are special immune cells that can control or regulate the body's immune response. We want to determine whether T regulatory cells are important participants in graft versus host disease (GVHD), infection and relapse. In GVHD, certain cells from the donated marrow or blood (the graft) attack the body of the transplant patient (the host). GVHD can affect many different parts of the body. The skin, eyes, stomach and intestines are affected most often. GVHD can range from mild to life-threatening. We do not know whether T regulatory cells can modify these conditions. We want to measure these T regulatory cells and learn if these cells do influence these conditions. If we learn that T regulatory cells do affect these conditions, then it may be possible to modify these cells for the benefit of transplant patients.

DETAILED DESCRIPTION:
To participate in this transplant, the patient will need to have a central line.

Before the transplant we will test the blood for viruses which can cause problems after the transplant. These viruses include Hepatitis B, cytomegalovirus and HIV. If the patient is positive for the AIDS virus, they will not be able to undertake the transplant.

Standard therapy: The patient will be given 6 doses of chemotherapy with a drug called Ara C in high doses (every 12 hours) which will begin 8 days before the stem cell transplant. Then, another chemotherapy drug called cyclophosphamide will be given in high doses by vein for two days on the 7th and 6th days before the transplant. A drug called MESNA will be given with cyclophosphamide. MESNA is used to decrease the side effects caused by cyclophosphamide. The patient will also receive an antibody called Campath (each day for 4 days before the transplant) to help destroy the immune system so that there is less host resistance to the growth of the donor cells. Radiation treatment will be given to the entire body on each day for 4 days before transplant. This will be given 2 times a day for 4 days. The chemotherapy and radiation treatment will last 8 days. If the patient has a diagnosis of T-cell Lymphoma, they will not be given the Ara-C.

Extra bone marrow tests may be recommended by the physician to check on the patients condition, especially if the marrow is slow to grow.

The day after the radiation treatment is completed; the patient will receive the healthy stem cells by vein. Once in the bloodstream, these stem cells will go to the bone marrow and should begin to grow.

In prevention of GvHD, the patient will also receive medicine called FK506 as well as low dose methotrexate. The FK506 will be given intravenously initially starting 2 days before the transplant and later by mouth (when they are able to take oral medications). This drug will be given each day for several weeks. Four doses of low dose methotrexate will be given intravenously. The methotrexate will be given on the day after the transplant, 3, 6 and 11 days after the transplant. If the GVHD cannot be controlled with FK506, other medicines may need to be given. The doctor will describe these medicines at that time.

Blood samples for research: To study how these cells are working in the patients system, blood samples will be taken each month for six months, at nine months, at one year, 2 years and 3 years following transplant. Approximately 6-8 teaspoons of blood will be collected each time. The total blood drawn for this study over three years should not exceed 1 and 3/4 cups. This amount is considered safe in adults. The amount of blood collected will be decreased in children and/or in patients where this amount of blood collection would not be appropriate.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with acute or chronic leukemia or advanced Hodgkin or non Hodgkin lymphoma or myelodysplastic/myeloproliferative disease who are unlikely to be cured by standard chemotherapy treatments. This includes patients who have relapsed after standard chemotherapy treatments and patients in first remission with unfavorable prognostic features.
* Using the standard 6 HLA antigen profile (HLA class I, A and B, and HLA class II, DRB1) a patient must have either a one HLA antigen mismatched related donor or an HLA matched or one antigen mismatched unrelated donor.

EXCLUSION CRITERIA:

* Patients with a life expectancy (less than or equal to 6 weeks) limited by disease other than leukemia.
* Patients with symptomatic cardiac failure unrelieved by medical therapy or evidence of significant cardiac dysfunction by echocardiogram (shortening fraction <20%).
* Patients with severe renal disease (i.e., creatinine greater than 3 times normal for age).
* Patients with pre-existing severe restrictive pulmonary disease (FVC less than 40% of predicted).
* Patients with severe hepatic disease (direct bilirubin greater than 3 mg/dl or AST greater than 500 IU/L).
* Patients with severe personality disorder or mental illness.
* Patients with severe infection that in the estimation of the principal investigator prohibits the use of ablative chemotherapy.
* Patients who are documented HIV positive.
* Patients with a Karnofsky performance score <70% or Lansky score <50%.

NOTE: Patients who would be excluded from treatment on this protocol strictly for laboratory abnormalities can be included at the principal investigator's discretion after consultation with the members of the SCT Policy and Procedures Committee.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krance, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Cohen JI, Jaffe ES, Dale JK, Pittaluga S, Heslop HE, Rooney CM, Gottschalk S, Bollard CM, Rao VK, Marques A, Burbelo PD, Turk SP, Fulton R, Wayne AS, Little RF, Cairo MS, El-Mallawany NK, Fowler D, Sportes C, Bishop MR, Wilson W, Straus SE. Characterization and treatment of chronic active Epstein-Barr virus disease: a 28-year experience in the United States. Blood. 2011 Jun 2;117(22):5835-49. doi: 10.1182/blood-2010-11-316745. Epub 2011 Mar 31. PMID 21454450

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stem Cell Transplant
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 24 patients were enrolled on the study and all of them received the conditioning treatment and the transplant.
Groups:
- Stem Cell Transplant: All patients will receive stem cell transplantation conditioning, GVHD prevention and stem cell infusion.
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (4.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Median Percentage of Treg Cells at 1 Year Post Transplant
Description: To define the biologic recovery and behavior of T regulatory cells for patients undergoing stem cell transplantation as specified in this protocol
Time Frame: 1 year
Population: Only 13 of the 24 patients enrolled were included in this analysis as only 13 patients have Treg values at 1 year.
Measure: Median (Inter-Quartile Range); unit: percentage of total CD4+ cells
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 13
percentage of total CD4+ cells | 6.9 [4.6 to 13.2]

ADVERSE EVENTS:
Arm/Group | Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 17/24
Other Adverse Events (participants affected / at risk) | 13/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Transplant (N=24)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 1 (1)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 1 (2)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (2)
Death (General disorders) | 1 (1) — Death not associated with CTCAE term - Multi-organ failure
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Bladder (urinary) (Infections and infestations) | 1 (1) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Bladder (urinary)
Infection with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 3 (4)
Infection with Grade 3 or 4 neutrophils - Bronchus (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
Infection - Other: Multiple viral infections (Infections and infestations) | 1 (1)
Infection - Other: Probable fungal disease (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Abdomen NOS (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 3 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 3 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper aerodigestive NOS (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 2 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
AST, SGOT (Metabolism and nutrition disorders) | 2 (2) — SGOT: serum glutamic oxaloacetic transaminase
Neurology - Other: Aseptic meningitis (Nervous system disorders) | 1 (1)
Neurology - Other: Cranial nerve VI palsy (Nervous system disorders) | 1 (1)
Neurology - Other: Peripheral neuropathy (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other: Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other: Respiratory distress: dyspnea + hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other: Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3)
Vascular - Other: Vaso Oclusive Disease (Vascular disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Transplant (N=24)
Hypotension (Cardiac disorders) | 2 (2)
PTT (Vascular disorders) | 2 (2) — PTT: Partial Thromboplastin Time
Diarrhea (Gastrointestinal disorders) | 2 (3)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 4 (5) — Two events were specified as oral cavity
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Infection - Other: CMV viremia (Infections and infestations) | 2 (2)
Infection with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 2 (2)
AST, SGOT (Metabolism and nutrition disorders) | 2 (2) — SGOT: serum glutamic oxaloacetic transaminase
Renal failure (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes